CLINICAL TRIAL: NCT07238088
Title: Monitoreo Activo de Mamografía y Orientación
Brief Title: Active Mammography and Counseling
Acronym: MAMO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Vivian Colon Lopez, Investigator Lead & Associate Director, University of Puerto Rico Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 2409000060; SUB-OTA No. 6922-03-COVID-S026 (Other Grant/Funding Number: WESTAT, INC.)
Record Dates: First submitted 2025-09-17; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Prevention
Keywords: breast cancer; Puerto Rico; cancer screening overdue; FQHC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study begins with a total of 1,020 participants, distributed equally across three intervention groups after filtering by municipality and applying inclusion criteria. Each group represents a progressively more intensive intervention level, designed to assess the impact of multi-component strategies on breast cancer screening rates among women aged 40-74 who are overdue for mammography by at least two years:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Educational Level (Experimental): Individual educational component
  Interventions: Behavioral: Individual Education
- Navigation Level (Experimental)
  Interventions: Behavioral: Individual Education; Other: Community Navigation
- Integration level (Experimental)
  Interventions: Behavioral: Individual Education; Other: Community Navigation; Other: Healthcare Providers Educational Intervention

INTERVENTIONS:
Behavioral: Individual Education — This component was developed using Intervention Mapping (IM) as a methodological framework and adapted from two evidence-based programs: "Unidas por la Vida" and "Nuestra Cocina: Mesa Buena, Vida Sana". The intervention includes one-on-one educational sessions led by Community Health Workers (CHWs), who will use tailored educational materials to guide participants and provide them with a take-home kit to promote and assist with mammography scheduling.
Other: Community Navigation — At this level, a community navigator service will be implemented to help participants overcome barriers to mammography screening. Seven community navigators will provide personalized support to address common challenges, including scheduling appointments, transportation, and access to healthcare services. These interventions leverage culturally tailored training to enable navigators to address barriers to breast cancer screening and enhance health literacy within their communities. The study intervention will include a specially designed training program for Community Navigators, emphasizing a culturally tailored curriculum to equip participants with the knowledge and skills necessary to educate and support their communities effectively.
  Arms: Integration level; Navigation Level
Other: Healthcare Providers Educational Intervention — The provider-level interventions will engage both clinical and administrative personnel who are actively employed at Federally Qualified Health Clinics (FQHCs). Two educational modules are being developed for the integration-level intervention. The educational content is designed to address provider-level barriers to breast cancer screening-an area that remains underexplored in the literature compared to patient-level factors. By engaging healthcare providers in FQHCs, this level aims to ensure women receive strong, consistent recommendations for mammography from trusted healthcare professionals.
  Arms: Integration level

SUMMARY:
The Puerto Rico Community Engagement Alliance (PR-CEAL) is an NIH-funded initiative which aims to improve health literacy and healthcare access across Puerto Rico. In 2024, the program developed a new study which goal is to improve breast cancer screening rates in Puerto Rico titled Monitoreo Activo de Mamografía y Orientación (MAMO). This multi-level study will recruit non-adherent women based on residence, age (40 to 74 years old), and having had two or more years since their last breast cancer screening. The intervention will focus on 39 municipalities with screening rates below the median, through three different levels: educational, navigation, and integration.

At the educational level, the intervention will employ a community-based recruitment strategy led by Community Health Workers (CHWs), who will identify eligible women at community venues and conduct follow-up via telephone to provide educational support. Drawing on findings from a previous pilot study and addressing barriers specific to non- adherent women, the navigation-level intervention will incorporate the role of a Community Navigator to deliver tailored support and facilitate breast cancer screening uptake through collaboration with local networks and partnerships. The integration-level intervention will build upon the educational and navigation components by enhancing knowledge, attitudes, skills, and organizational processes within Federally Qualified Health Clinics (FQHCs). This component is designed to foster a supportive healthcare environment that encourages routine mammography screening. The integration-level intervention will be implemented in four FQHCs across PR.

ELIGIBILITY:
Inclusion Criteria:

* Women (biological sex at birth) aged 40- 74
* Residing in one of 39 municipalities across Puerto Rico whose having a low breast cancer screening rate below the median (38.6%): Aibonito, Arecibo, Barceloneta, Caguas, Camuy, Comerío, Corozal, Florida, Las Piedras, Loíza, Naguabo, Vieques, Villalba, Añasco, Carolina, Cayey, Dorado, Guayanilla, Guaynabo, Isabela, Juana Diaz, Juncos, Luquillo, Manatí, Peñuelas, Quebradillas, Cabo Rojo, Canóvanas, Ceiba, Ciales, Coamo, Culebra, Fajardo, Morovis, Ponce, Sabana Grande, San Juan, Santa Isabel, and Trujillo Alto.
* Overdue for breast cancer screening by two or more years, in accordance with USPSTF guidelines
* Adequate cognitive orientation as verified by a brief version of the Mini-Mental State Examination
* Access to a telephone for follow-up and communication
* Ability to read and comprehend Spanish to engage with educational materials.

Exclusion Criteria:

* Women outside the specified age range (40-74)
* Up to date in breast cancer screening according to the USPSTF recommendations.
* No cognitive orientation
* Participants without access to a telephone
* Unable to read and comprehend Spanish
* Women undergoing active cancer treatment
* History of radical mastectomy

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants who self-reported having had a mammogram | Up to 12 months
  Participants will receive follow-up calls and emails every 3 months for one year to document their efforts to attend the clinic, undergo a mammogram, and receive a progress report from the clinicians about their mammogram result. The categories to collect this information are: Yes/No/Refuse to Answer.

SECONDARY OUTCOMES:
Changes in the mammogram rates considering intervention level: the Educational, Navigation, and Integration Levels | Up to 12 months
  The mammogram rate measure will be calculated based on the number of participants who reported undergoing a mammogram and receiving the results (numerator) with respect to the number of participants in the same intervention level (denominator). This measure will be collected at the intervention level.

OTHER OUTCOMES:
Changes in the patient-provider communication satisfaction considering intervention level: the Educational, Navigation, and Integration Levels | Up to 12 months
  Patient-provider communication satisfaction will be evaluated using a Likert Scale ranging from 0 (Strongly Agree) to 4 (Strongly Disagree). Through a phone call follow-up, the participant will provide their response. This measure will be collected at the intervention level.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Colon Lopez, PhD, MPH, Principal Investigator — UPR-Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided
According to our Data Management and Sharing Plan, raw data will only be available for study personnel and research activities included in the approved Institutional Review Board (IRB) protocol. To protect human research participants' privacy, rights, and confidentiality, we will manage all scientific data derived from human subjects in strict adherence to ethical guidelines and privacy protection measures, including de-identification techniques and obtaining Certificates of Confidentiality. The IRB will oversee all processes to guarantee compliance with these standards. Based on the statements, we will consider what data would be shared and for what purpose.